CLINICAL TRIAL: NCT03134157
Title: Evaluation the Effect of Simvastatin on Uterine Leiomyoma Development and Growth in Infertile Patients
Brief Title: The Effect of Simvastatin on Uterine Leiomyoma Development and Growth in Infertile Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Royan-Emb-029
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Infertility
Keywords: Leiomyoma simvastatin infertility
MeSH Terms: conditions — Infertility | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simvastatin and vaginal placebo (Experimental): The patients with leiomyoma receive simvastatin 40 mg orally+ vaginal placebo will be given every day for 3 months.
  Interventions: Drug: oral drug and vaginal placebo
- Simvastatin and oral placebo (Experimental): The patients with leiomyoma receive simvastatin 40 mg orally+ oral placebo will be given every day for 3 months.
  Interventions: Drug: oral drug and oral placebo
- Vaginal placebo+ oral placebo (Experimental): The patients with leiomyoma receive Vaginal placebo+ oral placebo every day for 3 months.
  Interventions: Drug: Vaginal placebo+ oral placebo

INTERVENTIONS:
Drug: oral drug and vaginal placebo — prescription of simvastatin 40 mg orally+ vaginal placebo every day for 3 months.
  Arms: Simvastatin and vaginal placebo
Drug: oral drug and oral placebo — prescription of simvastatin 40 mg orally+ oral placebo every day for 3 months.
  Arms: Simvastatin and oral placebo
Drug: Vaginal placebo+ oral placebo — prescription of Vaginal placebo + oral placebo every day for 3 months.
  Arms: Vaginal placebo+ oral placebo

SUMMARY:
Uterine leiomyomas with an estimated incidence of 50%-80% are the most common tumors of female reproductive system. Statins as a HMG-CoA reductase inhibitors inhibit the mevalonate pathway of cholesterol synthesis, thus have been known as a group of drugs used for treatment of hypercholesterolemia. Statins inhibit proliferation of several cell types including vascular smooth muscle, hepatocytes and other cell types. Leiomyomas are benign uterine tumors characterized by smooth muscle proliferation and excessive deposition of extracellular matrix. In the present study we aim to evaluate the effect of simvastatin on uterine leiomyoma development and growth.

DETAILED DESCRIPTION:
The proposal of the present study approved by our institutional review boards and institution's ethical committee, and all participants will sign a written consent before enter to study. All patients will be randomly divided into three groups and will be randomized to receive simvastatin 40 mg orally + vaginal placebo, simvastatin 40 mg vaginally + oral placebo and vaginal placebo + oral placebo for 3 months.

CBC, Lipid profile, kidney & Liver function tests, FBS & hormonal evaluation will be performed before and after the treatment. Ultrasound examination will be performed before and after the treatment for determining of the number, size, and site of the myoma and also size of the uterus.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years
* Intramural Fibroids confirmed by ultrasound
* Presence of at least one fibroid with size >4 cm or two fibroids with size >3 cm detected by pelvic ultrasound.
* Presence of at least 3 fibroids with size <3 cm and a history of 2 IVF failures.
* Number of fibroids ≤ 5
* BMI>25 Kg/m2

Exclusion Criteria:

* Pregnancy
* Hormonal contraception or any hormonal therapy received in the last 3 months
* Alcohol consumption
* Allergic to simvastatin
* Suspicion or diagnosis of cancer
* Signs or symptoms of mental illness, hepatic dysfunction, myopathic syndromes, diabetes mellitus, renal disease, Cardiovascular disease, hypothyroidism, hypotension, neuropathy, lupus and cataract
* Hb ≤ 7
* Taking antifungal medications, Lipid-Lowering medications (gemfibrozil, clofibrate), warfarin, danazol and erythromycin in the last one month.
* Severe male factor
* Severe endometriosis
* Diminished ovarian reserve

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-09-14 (Estimated)

PRIMARY OUTCOMES:
Uterine fibroid size | 3 months
  Evaluation the size of Uterine fibroid withultrasound.

SECONDARY OUTCOMES:
Uterine size | 3months
  Evaluation the uterine size with ultrasound.
Plasma concentration of Vitamin D3 | 3 months
  Evaluation the Plasma concentration of Vitamin D3 with blood sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Ashrafi, MD, Study Director — ) Endocrinology and Female Infertility Department, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Firoozeh Ahmadi, MD, Study Director — ) Endocrinology and Female Infertility Department, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Nadia Jahangiri, MSc, Principal Investigator — ) Endocrinology and Female Infertility Department, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehrān, Iran

IPD SHARING:
Plan to Share IPD: No